CLINICAL TRIAL: NCT04510012
Title: Characterizing the Immune Response and Neuronal Damage in SARS-CoV-2 Infected Individuals
Brief Title: Characterizing the Immune Response and Neuronal Damage in COVID-19
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Other Study IDs: nCOV19
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: SARS-CoV Infection; Covid-19
Keywords: Innate immune response; Adaptive immune response; Inflammation; Neurological damage
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; COVID-19; Inflammation; Trauma, Nervous System | interventions — Adaptive Immunity; Complement Activation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Plasma, Peripheral Blood Mononuclear Cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Mild COVID-19: SARS-Cov-2 infected individuals with mild symptoms (WHO Ordinal Scale for Clinical Improvement in COVID-19: scores 1-2)
  Interventions: Other: Analysis of cytokine response, innate and adaptive immune response, complement activation, and serum neurofilaments as a marker of neurological damage.
- Moderate COVID-19: SARS-Cov-2 infected individuals with moderate symptoms (WHO Ordinal Scale for Clinical Improvement in COVID-19: scores 3-4)
  Interventions: Other: Analysis of cytokine response, innate and adaptive immune response, complement activation, and serum neurofilaments as a marker of neurological damage.
- Severe COVID-19: SARS-Cov-2 infected individuals with severe symptoms (WHO Ordinal Scale for Clinical Improvement in COVID-19: scores 5-8)
  Interventions: Other: Analysis of cytokine response, innate and adaptive immune response, complement activation, and serum neurofilaments as a marker of neurological damage.

INTERVENTIONS:
Other: Analysis of cytokine response, innate and adaptive immune response, complement activation, and serum neurofilaments as a marker of neurological damage. — Analysis of cytokine response, innate and adaptive immune response, complement activation, and serum neurofilaments as a marker of neurological damage.

SUMMARY:
The Investigators plan to study the innate and adaptive immune response, the inflammatory response, and associated complications such as complement activation and neurological damage in SARS-Cov-2 infected individuals. Patients with mild, moderate and severe COVID-19 disease will be enrolled.

DETAILED DESCRIPTION:
The severity of coronavirus disease 2019 (COVID-19) ranges from asymptomatic infection to severe illness requiring mechanical ventilation. Immunological factors which lead to severe disease in certain COVID-19 patients remain incompletely understood. Neurological damage and complement activation may be a consequence of excess inflammation in severe COVID-19. The investigators plan to study the innate and adaptive immune response and potentially associated complications such as neurological damage and complement activation in mild, moderate and severe COVID-19 courses.

ELIGIBILITY:
Inclusion Criteria:

* PCR confirmed SARS-Cov-2 infection

Exclusion Criteria:

* Refusal to participate
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (≤ 18 years) patients with PCR confirmed SARS-Cov-2 infection
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2020-03-05 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Cytokine response to SARS-Cov-2 | At enrollment
  Measurement of cytokine concentration (pg/ml) in serum (IL-6, IL-8, IL-1b,TNF-alpha)
Cytokine response to SARS-Cov-2 | 28 days (+/-7) after enrollment
  Measurement of cytokine concentration (pg/ml) in serum (IL-6, IL-8, IL-1b,TNF-alpha)
Innate immune response to SARS-Cov-2 | At enrollment
  Measurement of HLA-DR expression on CD14+ cells (flowcytometry)
Innate immune response to SARS-Cov-2 | 3 days after enrollment
  Measurement of HLA-DR expression on CD14+ cells (flowcytometry)
Innate immune response to SARS-Cov-2 | 5 days after enrollment
  Measurement of HLA-DR expression on CD14+ cells (flowcytometry)
Humoral immune response | At enrollment
  Measurement of neutralizing SARS-Cov-2 antibody concentrations (plaque reduction assay)
Cell mediated immune response | At enrollment
  Measurement of frequencies of SARS-Cov-2 specific T-cells (ELISPOT assay)
Cell mediated immune response | 28 days (+/-7) after enrollment
  Measurement of frequencies of SARS-Cov-2 specific T-cells (ELISPOT assay)
Neurological damage | At enrollment
  Measurement of neurofilament light chains in serum (on ELLA platform; Protein Simple, Bio-techne)
Neurological damage | 28 days (+/-7) after enrollment
  Measurement of neurofilament light chains in serum (on ELLA platform; Protein Simple, Bio-techne)

SECONDARY OUTCOMES:
Complement activation | At enrollment
  Measurement of factor B, factor H, factor I, C3a, C4a, C5a, SC5b9
Complement activation | 28 days (+/-7) after enrollment
  Measurement of factor B, factor H, factor I, C3a, C4a, C5a, SC5b9

CONTACTS AND LOCATIONS:
Overall Officials: Cédric Hirzel, MD, Principal Investigator — Department of Infectious Diseases, Bern University Hospital, Bern, Switzerland; Leib L Stephen, MD, Principal Investigator — Institute for Infectious Diseases; Bern University; Jörg C Schefold, MD, Principal Investigator — Department of Intensive Care Medicine, Inselspital, Bern University Hospital, University of Bern, Switzerland
Locations (1):
- Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ruggeri T, De Wit Y, Scharz N, van Mierlo G, Angelillo-Scherrer A, Brodard J, Schefold JC, Hirzel C, Jongerius I, Zeerleder S. Immunothrombosis and Complement Activation Contribute to Disease Severity and Adverse Outcome in COVID-19. J Innate Immun. 2023;15(1):850-864. doi: 10.1159/000533339. Epub 2023 Nov 8. PMID 37939687